CLINICAL TRIAL: NCT05586906
Title: Noninvasive Early Detection of Lung Allograft Dysfunction After Lung Transplantation With Multiple Breath Washout Test: Lung Clearance Index as an Early Marker
Brief Title: Noninvasive Early Detection of Lung Allograft Dysfunction After Lung Transplantation With Multiple Breath Washout Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ilhan Inci, Prof. Dr., University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01610
Record Dates: First submitted 2017-11-02; First posted 2022-10-19 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chronic Rejection of Lung Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Multiple Breath Washout (MBW) tests — LCI measurements (EXHALYZER® D with Nitrogen Washout System, ECO Medics AG) will be performed every month during follow-up beginning 3 months after lung transplantation.

SUMMARY:
Chronic rejection, more commonly called bronchiolitis obliterans syndrome (BOS), is the leading cause of death beyond the first year post lung transplantation. The diagnosis of BOS is typically made by clinical, physiological, and radiographic parameters. Early detection would be desirable since it allows treatment modification to stop or delay the process. In the last few years there has been a growing interest in lung clearance index (LCI), a measure of lung physiology derived from multiple breath washout tests. LCI is derived from Multiple Breath Washout (MBW) tests. Early detection of BOS with LCI measurement will allow the investigators early recognition of this chronic rejection form and with early institution of the enhanced treatment survival will increase. All paticipants who underwent bilateral lung transplantation at Zurich University Hospital will be included. The measurement will be done 3 months after lung transplantation. Approximately 90 paticipants will be included. The follow-up will be 5 years. If the investigators could detect the development of BOS with this novel method before the clinical deterioration (fall in lung function) the investigators can start the available treatment options before irreversible damage occurs. This might increase overall survival in the study cohort.

DETAILED DESCRIPTION:
Lung transplantation is a treatment option for patients with advanced lung disease or irreversible pulmonary failure. Despite advancements in surgical techniques, lung preservation, immunosuppression, and management of ischemia/reperfusion injury and infections, chronic allograft rejection continue to be a major problem. Chronic rejection, more commonly called bronchiolitis obliterans syndrome (BOS), is the leading cause of death beyond the first year post lung transplantation.

BOS affects 50% or more of recipients who survive beyond 5 years and accounts for a considerable proportion of cases of lung allograft loss and recipient death beyond 3 months post-transplant. It is the leading cause of death for recipients who survive beyond 1 year post-transplant, and it is widely perceived as the physiological surrogate of immunologically-mediated phenomena due to many observations that include its association with acute cellular rejection, the tendency of recipients who develop BOS to have greater degrees of human leukocyte antigen mismatch, and accumulating evidence of the involvement of autoimmune pathways. Furthermore, there are striking similarities to obliterative bronchiolitis that can occur in allogeneic bone marrow or stem cell transplant recipients as well as in patients with connective tissue diseases, which are also perceived as alloimmune or autoimmune disorders, respectively. Therefore, BOS is frequently equated with the term chronic rejection.

The diagnosis of BOS is typically made by clinical, physiological, and radiographic parameters. Early detection would be desirable since it allows treatment modification to stop or delay the process. Due to the sporadic or patchy involvement of obliterative bronchiolitis, pathologic diagnosis can be missed by transbronchial biopsies (TBB), which are often performed to exclude other diagnoses including acute rejection or infection. Histologically, early lesions of BOS demonstrate partial or complete obstruction of the small airways.

Currently, radiographic imaging is not used as a diagnostic tool in transplant recipients when evaluating for BOS; however, high resolution computed tomography (HRCT) imaging with inspiratory and expiratory views may be helpful when considering the diagnosis.

In the last few years there has been a growing interest in lung clearance index (LCI), a measure of lung physiology derived from multiple breath washout tests. LCI is derived from Multiple Breath Washout (MBW) tests. The test involves following the washout of an inert tracer gas from the lungs during relaxed tidal breathing. The tracer gas can be nitrogen that is normally resident in the lungs, washed out when the participant is switched to breathing 100% oxygen.

This test (lung clearing index) detects early airways disease in children, and is more sensitive and easier to perform in this population than conventional lung function tests. With an appreciation of the importance of earlier identification of airways dysfunction, and prevention of irreversible structural airway changes, methods of following airways disease in these ''silent years'' are especially important. LCI has now been reported in studies involving all age groups, from infants to adults, and has a narrow range of normal over this wide age range, making it especially suitable for long-term follow-up studies.

Specific Aim:

Early detection of development BOS with LCI before deterioration in the conventional lung function test occurs.

Hypothesis:

Early detection of BOS with LCI measurement will allow the investigators early recognition of this chronic rejection form and with early institution of the enhanced treatment survival will increase.

Study population:

All participants who underwent bilateral lung transplantation at Zurich University Hospital will be included. The measurement will be done 3 months after lung transplantation. Approximately 90 patients will be included. The follow-up will be 5 years.

Method:

LCI measurements (EXHALYZER® D with Nitrogen Washout System, ECO Medics AG) will be performed every month during follow-up beginning 3 months after lung transplantation. The test will be repeated every month. Follow-up will be 5 years. Individually the follow-up period might be prolonged.

Relevance and impact:

If the investigators could detect the development of BOS with this novel method before the clinical deterioration (fall in lung function) the investigators can start the available treatment options before irreversible damage occurs. This might increase overall survival in study cohort.

ELIGIBILITY:
Inclusion Criteria:

* All recipients who underwent bilateral lung transplantation at Zurich University Hospital will be included.

Exclusion Criteria:

* Retransplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Lung Clearance Index (LCI) derived from Multiple Breath Washout Test (MBWT) | 5 years
  LCI 2.5 (ext): lung clearance index at normalised end tidal concentration of N2 2.5% extrapolated
FEV1 (L) | 5 years
  Forced expiratory volume in one second measured in liters
FEV1 (%) | 5 years
  percent of forced expiratory volume in one second measured in percent

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Steinack, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland